CLINICAL TRIAL: NCT01396447
Title: A Double-Blind, Placebo-Controlled Evaluation of the Safety and Efficacy of Cariprazine in Patients With Bipolar Depression
Brief Title: Safety, Tolerability, and Efficacy of Cariprazine in Participants With Bipolar Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Gedeon Richter Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RGH-MD-56; 2011-002334-39 (EudraCT Number)
Record Dates: First submitted 2011-07-15; First posted 2011-07-18 (Estimated); Results first posted 2018-05-01 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-03

CONDITIONS: Depression, Bipolar
Keywords: Bipolar I disorder; Bipolar depression; Depression; Bipolar disorder
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — cariprazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Participants received placebo orally once a day for 8 weeks.
  Interventions: Drug: Placebo
- Cariprazine 0.75 mg (Experimental): Participants received cariprazine 0.5 mg orally once on Days 1-2 and cariprazine 0.75 mg orally once a day starting on Day 3 for the remainder of the 8 week treatment period.
  Interventions: Drug: Cariprazine
- Cariprazine 1.5 mg (Experimental): Participants received cariprazine 0.5 mg orally once on Days 1-2, cariprazine 0.75 mg orally once on Days 3-4, cariprazine 1.0 mg orally once on Days 5-7, and cariprazine 1.5 mg orally once a day starting on Day 8 for the remainder of the 8 week treatment period.
  Interventions: Drug: Cariprazine
- Cariprazine 3.0 mg (Experimental): Participants received cariprazine 0.5 mg orally once on Days 1-2, cariprazine 0.75 mg orally once on Days 3-4, cariprazine 1.0 mg orally once on Days 5-7, cariprazine 1.5 mg orally on Days 8-14, and cariprazine 3.0 mg orally once a day starting on Day 15 for the remainder of the 8 week treatment period.
  Interventions: Drug: Cariprazine

INTERVENTIONS:
Drug: Placebo — Placebo was supplied in capsules.
  Arms: Placebo
Drug: Cariprazine — Cariprazine was supplied in capsules.
  Arms: Cariprazine 0.75 mg; Cariprazine 1.5 mg; Cariprazine 3.0 mg

SUMMARY:
The objective of this study was to evaluate the efficacy, safety, and tolerability of cariprazine relative to placebo for the treatment of participants with bipolar depression.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have provided informed consent prior to any study specific procedures.
* Participants currently meeting the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria for bipolar I disorder as confirmed by the Structured Clinical Interview (SCID) with a current with a current major depressive episode of at least 4 weeks and not exceeding 12 months in duration.
* Participants with normal physical examination, laboratory, vital signs, and/or echocardiogram (ECG).
* Verified previous manic or mixed episode.
* Participants with a total Hamilton Rating Scale for Depression (HAMD)-17 score ≥ 20.
* Participants with a HAMD-17 item 1 score ≥ 2.
* Participants with a Clinical Global Impression of Severity (CGI-S) score ≥ 4.

Exclusion Criteria:

* Participants with a DSM-IV-TR diagnosis of an axis I disorder other than bipolar I disorder that was the primary focus of treatment within the previous 6 months.
* Women who are pregnant or breast feeding
* Participants with Young Mania Rating Scale (YMRS) total score > 10
* Participants who have dementia, mental retardation, schizophrenia/schizoaffective disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 584 (Actual)
Dates: Start 2011-07-26 (Actual); Primary Completion 2014-01-10 (Actual); Study Completion 2014-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Willie Earley, MD, Study Director — Allergan
Locations (88):
- United States (38):
  - Forest Investigative Site 021, Birmingham, Alabama
  - Forest Investigative Site 017, Springdale, Arkansas
  - Forest Investigative Site 030, Beverly Hills, California
  - Forest Investigative Site 018, Cerritos, California
  - Forest Investigative Site 028, Costa Mesa, California
  - Forest Investigative Site 015, Oceanside, California
  - Forest Investigative Site 011, Temecula, California
  - Forest Investigative Site 012, Jacksonville, Florida
  - Forest Investigative Site 035, Orlando, Florida
  - Forest Investigative Site 013, Winter Park, Florida
  - Forest Investigative Site 038, Atlanta, Georgia
  - Forest Investigative Site 005, Atlanta, Georgia
  - Forest Investigative Site 029, Chicago, Illinois
  - Forest Investigative Site 024, Indianapolis, Indiana
  - Forest Investigative Site 031, Prairie Village, Kansas
  - Forest Investigative Site 041, Lake Charles, Louisiana
  - Forest Investigative Site 040, Shreveport, Louisiana
  - Forest Investigative Site 039, Flowood, Mississippi
  - Forest Investigative Site 026, Creve Coeur, Missouri
  - Forest Investigative Site 037, Las Vegas, Nevada
  - Forest Investigative Site 023, Cherry Hill, New Jersey
  - Forest Investigative Site 014, Marlton, New Jersey
  - Forest Investigative Site 006, Albuquerque, New Mexico
  - Forest Investigative Site 003, Brooklyn, New York
  - Forest Investigative Site 025, New York, New York
  - Forest Investigative Site 036, Canton, Ohio
  - Forest Investigative Site 008, Dayton, Ohio
  - Forest Investigative Site 042, Salem, Oregon
  - Forest Investigative Site 009, Allentown, Pennsylvania
  - Forest Investigative Site 010, Media, Pennsylvania
  - Forest Investigative Site 033, Lincoln, Rhode Island
  - Forest Investigative Site 019, Memphis, Tennessee
  - Forest Investigative Site 007, Dallas, Texas
  - Forest Investigative Site 016, Houston, Texas
  - Forest Investigative Site 027, Houston, Texas
  - Forest Investigative Site 020, San Antonio, Texas
  - Forest Investigative Site 043, Bellevue, Washington
  - Forest Investigative Site 032, Seattle, Washington
- Bulgaria (11):
  - Forest Investigative Site 311, Kardzhali
  - Forest Investigative Site 307, Kazanlak
  - Forest Investigative Site 310, Lovech
  - Forest Investigative Site 313, Novi Iskar
  - Forest Investigative Site 309, Pazardzhik
  - Forest Investigative Site 302, Pleven
  - Forest Investigative Site 301, Plovdiv
  - Forest Investigative Site 305, Sofia
  - Forest Investigative Site 306, Sofia
  - Forest Investigative Site 308, Tsarev Brod
  - Forest Investigative Site 312, Tserova Koria
- Canada (3):
  - Forest Investigative Site 102, Kelowna, British Columbia
  - Forest Investigative Site 103, Penticton, British Columbia
  - Forest Investigative Site 101, Chatham, Ontario
- Colombia (6):
  - Forest Investigative Site 804, Barranquilla
  - Forest Investigative Site 806, Barranquilla
  - Forest Investigative Site 803, Bogotá
  - Forest Investigative Site 805, Bogotá
  - Forest Investigative Site 808, Bogotá
  - Forest Investigative Site 807, Pereira
- Russia (18):
  - Forest Investigative Site 601, Arkhangelsk
  - Forest Investigative Site 605, Moscow
  - Forest Investigative Site 607, Moscow
  - Forest Investigative Site 611, Moscow
  - Forest Investigative Site 619, Moscow
  - Forest Investigative Site 603, Nizhny Novgorod
  - Forest Investigative Site 604, Saint Petersburg
  - Forest Investigative Site 606, Saint Petersburg
  - Forest Investigative Site 602, Saint Petersburg
  - Forest Investigative Site 613, Saint Petersburg
  - Forest Investigative Site 608, Saint Petersburg
  - Forest Investigative Site 615, Saint Petersburg
  - Forest Investigative Site 612, Saint Petersburg
  - Forest Investigative Site 617, Samara
  - Forest Investigative Site 616, Saratov
  - Forest Investigative Site 609, Tomsk
  - Forest Investigative Site 618, Tver'
  - Forest Investigative Site 610, Voronezh
- Ukraine (12):
  - Forest Investigative Site 707, Kerch, AR Crimea
  - Forest Investigative Site 709, Kherson, Vil. Stepanivka
  - Forest Investigative Site 714, Donetsk
  - Forest Investigative Site 712, Ivano-Frankivsk
  - Forest Investigative Site 703, Kharkiv
  - Forest Investigative Site 704, Kharkiv
  - Forest Investigative Site 702, Kharkiv
  - Forest Investigative Site 708, Kyiv
  - Forest Investigative Site 701, Kyiv
  - Forest Investigative Site 710, Odesa
  - Forest Investigative Site 706, Simferopol
  - Forest Investigative Site 705, Vinnytsia

REFERENCES:
- [Derived] McIntyre RS, Llorca PM, Aronin LC, Yu J, Nguyen HB. Effect of Cariprazine on Anhedonia in Patients with Bipolar I Depression: Post Hoc Analysis of Three Randomized Placebo-Controlled Clinical Trials. Adv Ther. 2025 Jan;42(1):246-260. doi: 10.1007/s12325-024-03009-2. Epub 2024 Nov 9. PMID 39520655
- [Derived] Vieta E, Calabrese JR, Whelan J, Tohen M, Earley WR. The efficacy of cariprazine on function in patients with bipolar depression: a post hoc analysis of a randomized controlled trial. Curr Med Res Opin. 2021 Sep;37(9):1635-1643. doi: 10.1080/03007995.2021.1932446. Epub 2021 Jun 7. PMID 34034612
- [Derived] Citrome L, Yatham LN, Patel MD, Barabassy A, Hankinson A, Earley WR. Cariprazine and akathisia, restlessness, and extrapyramidal symptoms in patients with bipolar depression. J Affect Disord. 2021 Jun 1;288:191-198. doi: 10.1016/j.jad.2021.03.076. Epub 2021 Mar 31. PMID 33915374
- [Derived] Thase ME, Harrington A, Calabrese J, Montgomery S, Niu X, Patel MD. Evaluation of MADRS severity thresholds in patients with bipolar depression. J Affect Disord. 2021 May 1;286:58-63. doi: 10.1016/j.jad.2021.02.043. Epub 2021 Feb 20. PMID 33677183
- [Derived] Yatham LN, Vieta E, McIntyre RS, Jain R, Patel M, Earley W. Broad Efficacy of Cariprazine on Depressive Symptoms in Bipolar Disorder and the Clinical Implications. Prim Care Companion CNS Disord. 2020 Sep 17;22(5):20m02611. doi: 10.4088/PCC.20m02611. PMID 32942346
- [Derived] Earley WR, Burgess M, Rekeda L, Hankinson A, McIntyre RS, Suppes T, Calabrese JR, Yatham LN. A pooled post hoc analysis evaluating the safety and tolerability of cariprazine in bipolar depression. J Affect Disord. 2020 Feb 15;263:386-395. doi: 10.1016/j.jad.2019.11.098. Epub 2019 Nov 22. PMID 31969269
- [Derived] Durgam S, Earley W, Lipschitz A, Guo H, Laszlovszky I, Nemeth G, Vieta E, Calabrese JR, Yatham LN. An 8-Week Randomized, Double-Blind, Placebo-Controlled Evaluation of the Safety and Efficacy of Cariprazine in Patients With Bipolar I Depression. Am J Psychiatry. 2016 Mar 1;173(3):271-81. doi: 10.1176/appi.ajp.2015.15020164. Epub 2015 Nov 6. PMID 26541814

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants with a diagnosis of bipolar I disorder with a current major depressive episode were considered for participation in the study.
Period: Overall Study
Arm/Group | Placebo | Cariprazine 0.75 mg | Cariprazine 1.5 mg | Cariprazine 3.0 mg
Started | 148 | 143 | 147 | 146
Received Treatment | 145 | 141 | 146 | 146
Completed | 105 | 103 | 117 | 94
Not Completed | 43 | 40 | 30 | 52
Not completed — Did Not Receive Treatment | 3 | 2 | 1 | 0
Not completed — Adverse Event | 15 | 12 | 12 | 17
Not completed — Insufficient Therapeutic Response | 5 | 5 | 2 | 4
Not completed — Protocol Violation | 5 | 2 | 3 | 7
Not completed — Withdrawal of Consent | 11 | 9 | 4 | 15
Not completed — Lost to Follow-up | 4 | 8 | 7 | 9
Not completed — Other Miscellaneous Reasons | 0 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population: All randomized participants who received at least 1 dose of investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Cariprazine 0.75 mg | Cariprazine 1.5 mg | Cariprazine 3.0 mg | Total
Number analyzed (Participants) | 145 | 141 | 146 | 146 | 578
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (12.0) | 40.1 (11.2) | 40.9 (11.4) | 42.8 (10.8) | 41.9 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 91 | 92 | 88 | 360
  Male | 56 | 50 | 54 | 58 | 218
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 13 | 11 | 12 | 48
  Not Hispanic or Latino | 133 | 128 | 135 | 134 | 530
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 110 | 111 | 109 | 113 | 443
  Black or African-American | 30 | 26 | 30 | 26 | 112
  Asian | 1 | 1 | 2 | 0 | 4
  American Indian or Alaska Native | 2 | 1 | 1 | 3 | 7
  Other | 2 | 2 | 4 | 4 | 12
Weight [Mean (Standard Deviation); unit: kg] | 79.98 (17.08) | 80.81 (18.36) | 81.43 (16.79) | 81.45 (17.86) | 80.92 (17.49)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.81 (5.27) | 28.42 (5.71) | 28.44 (5.39) | 28.28 (5.64) | 28.24 (5.50)
Waist circumference [Mean (Standard Deviation); unit: cm] | 91.40 (14.24) | 93.32 (15.45) | 93.38 (14.55) | 93.24 (15.40) | 92.83 (14.90)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Montgomery-Åsberg Depression Rating Scale Total Score at Week 6
Description: The Montgomery-Åsberg Depression Rating Scale is a 10-item, clinician-rated scale that evaluates the participant's depressive symptomatology during the past week. Participants are rated on items assessing feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty in concentration, and lack of interest. Each item is scored on a 7-point scale with a score of 0 reflecting no symptoms and a score of 6 reflecting symptoms of maximum severity. The scores on the 10 items are summed for a total score that can range from 0 to 60. A higher score indicates greater depression. A negative change score indicates improvement.
Time Frame: Baseline to Week 6
Population: Intent-to-treat population: All randomized participants who took at least 1 dose of investigational product and had at least 1 post-Baseline assessment of the Montgomery-Åsberg Depression Rating Scale.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Cariprazine 0.75 mg | Cariprazine 1.5 mg | Cariprazine 3.0 mg
Number analyzed (Participants) | 141 | 140 | 145 | 145
units on a scale | -11.1 (0.9) | -13.0 (0.9) | -15.1 (0.8) | -13.7 (0.9)
Statistical Analysis 1: Comparison: Placebo vs Cariprazine 0.75 mg; Test type: Superiority; p = 0.1292, Repeated measures mixed-effects model — The analysis included treatment group, pooled study center, visit, and treatment-group-by-visit interaction as fixed effects and the baseline value and baseline value-by-visit interaction as covariates; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-4.3 to 0.5] — Cariprazine 0.75 mg vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Cariprazine 1.5 mg; Test type: Superiority; p = 0.0010, Repeated measures mixed-effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.0, 95% CI 2-sided [-6.3 to -1.6] — Cariprazine 1.5 mg vs Placebo
Statistical Analysis 3: Comparison: Placebo vs Cariprazine 3.0 mg; Test type: Superiority; p = 0.0374, Repeated measures mixed-effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-4.9 to -0.1] — Cariprazine 3.0 mg vs Placebo

2. Secondary Outcome: Change From Baseline in the Clinical Global Impressions-Severity Total Score at Week 6
Description: The Clinical Global Impressions-Severity scale is a clinician-rated scale that measures the overall severity of a participant's illness in comparison with the severity of illness in other participants the physician has observed. The participant is rated on a scale from 1 to 7 with 1 indicating a "normal state" and 7 indicating "among the most extremely ill participants." A higher score indicates greater illness. A negative change score indicates improvement.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Cariprazine 0.75 mg | Cariprazine 1.5 mg | Cariprazine 3.0 mg
Number analyzed (Participants) | 141 | 140 | 145 | 145
units on a scale | -1.0 (0.1) | -1.1 (0.1) | -1.4 (0.1) | -1.3 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Cariprazine 0.75 mg; The analysis included treatment group, pooled study center, visit, and treatment-group-by-visit interaction as fixed effects and the baseline value and baseline value-by-visit interaction as covariates; Test type: Superiority; p = 0.3025, Repeated measures mixed-effects model; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.4 to 0.1] — Cariprazine 0.75 mg vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Cariprazine 1.5 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0044, Repeated measures mixed-effects model; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.6 to -0.2] — Cariprazine 1.5 mg vs Placebo
Statistical Analysis 3: Comparison: Placebo vs Cariprazine 3.0 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0489, Repeated measures mixed-effects model; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.5 to -0.0] — Cariprazine 3.0 mg vs Placebo

ADVERSE EVENTS:
Time Frame: Adverse Events were collected and recorded from the time the participant signs the informed consent form until 30 days after the last dose of treatment.
Description: Safety population: All randomized participants who took at least 1 dose of investigational product.
Arm/Group | Placebo | Cariprazine 0.75 mg | Cariprazine 1.5 mg | Cariprazine 3.0 mg
All-Cause Mortality (participants affected / at risk) | 0/145 | 0/141 | 0/146 | 0/146
Serious Adverse Events (participants affected / at risk) | 5/145 | 1/141 | 2/146 | 2/146
Other Adverse Events (participants affected / at risk) | 42/145 | 43/141 | 51/146 | 56/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=145) | Cariprazine 0.75 mg (N=141) | Cariprazine 1.5 mg (N=146) | Cariprazine 3.0 mg (N=146)
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Vertigo CNS origin (Nervous system disorders) | 0 | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0 | 0
Hypomania (Psychiatric disorders) | 0 | 0 | 1 | 0
Mania (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=145) | Cariprazine 0.75 mg (N=141) | Cariprazine 1.5 mg (N=146) | Cariprazine 3.0 mg (N=146)
Nausea (Gastrointestinal disorders) | 7 | 12 | 12 | 12
Diarrhoea (Gastrointestinal disorders) | 10 | 2 | 9 | 3
Akathisia (Nervous system disorders) | 2 | 4 | 7 | 21
Headache (Nervous system disorders) | 17 | 11 | 11 | 10
Somnolence (Nervous system disorders) | 7 | 6 | 10 | 10
Insomnia (Psychiatric disorders) | 12 | 16 | 10 | 17
Restlessness (Psychiatric disorders) | 5 | 4 | 4 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study. Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.